CLINICAL TRIAL: NCT03779958
Title: Alternatives to Hand Therapy for Hand Surgery Patients
Status: Withdrawn | Type: Observational
Why Stopped: Logistics (Research Staffing)
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Other Study IDs: 47777
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Carpal Tunnel Syndrome; Trigger Finger; Ganglion Cysts; Distal Radius Fracture; Finger Fracture; De Quervain Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome; Trigger Finger Disorder; Ganglion Cysts; Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: All patients will be given information about a mobile app to use during the recovery period to assist with hand therapy activities
  Interventions: Other: Mobile App

INTERVENTIONS:
Other: Mobile App — a mobile app that demonstrates hand therapy exercises

SUMMARY:
Patients will be asked to use a mobile phone app to conduct their hand therapy after having hand surgery.

DETAILED DESCRIPTION:
Patients who are undergoing the included procedures will be informed of the study & consented. They will be given information on how to download the app & input their surgery date. The app will guide the patient through various hand therapy exercises and ask them to record their QuickDASH, PSFS and VAS Pain weekly.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing the following procedures: carpal tunnel release, trigger finger release, distal radius fracture fixation, de quervains release, cyst excision, finger fracture fixation
* smart phone that is compatible with the app

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting to a single hand surgery clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
QuickDASH | once a week for 6 weeks
  The QD is a short form of the DASH, which measures disability of the arm, shoulder and hand. it is scored 0-100, with higher scores indicating higher disability

SECONDARY OUTCOMES:
Patient Specific Functional Scale | once a week for 6 weeks
  the PSFS is a validated measure of disability, that is scored on a 0-10 scale with lower scored indicating higher disability.
VAS Pain | once a week for 6 weeks
  VAS pain is a validated measure of pain, scored 0-10, with higher scores indicating higher pain

CONTACTS AND LOCATIONS:
Overall Officials: Robin N Kamal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No